CLINICAL TRIAL: NCT06820489
Title: A Three-arm Randomized Controlled Trial Comparing Transmucosal Augmentation Techniques in Immediate Implant Placement
Brief Title: Comparison of Three Transmucosal Augmentation Techniques in Immediate Implant Placement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONZ-2024-0529
Record Dates: First submitted 2025-02-05; First posted 2025-02-11 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Bone Resorption
Keywords: Dental Implant, Single-Tooth; Immediate; Connective tissue graft
MeSH Terms: conditions — Bone Resorption

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: As this RCT concerns a surgical intervention, patients and treating clinicians can not be masked.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional connective tissue graft (Active Comparator): Connective tissue graft immediately inserted in buccal pouch
  Interventions: Procedure: Conventional connective tissue graft after immediate implant placement
- Scarf connective tissue graft (Experimental): Connective tissue graft immediately fixed onto the buccal mucosa.
  Interventions: Procedure: Scarf connective tissue graft after immediate implant placement
- Dual zone concept (Experimental): Bone material condensed up to the buccal soft tissue margin.
  Interventions: Procedure: Dual zone concept after immediate implant placement

INTERVENTIONS:
Procedure: Conventional connective tissue graft after immediate implant placement — A pouch is made in the buccal mucosa extending 3 mm below the buccal bone crest. Thereupon, a free gingival graft is harvested from the palatal mucosa and de-epithelialized. The CTG is brought into the pouch and fixed with two single sutures onto the buccal mucosa. A healing abutment is installed, which is replaced by a provisional implant crown 2 days later. Sutures are removed 1 week after the surgery.
  Arms: Conventional connective tissue graft
Procedure: Scarf connective tissue graft after immediate implant placement — No pouch is made in the recipient site. A free gingival graft is harvested from the palatal mucosa and de-epithelialized. The small CTG is fixed at the transmucosal aspect onto the buccal mucosa. A healing abutment is installed, which is replaced by a provisional implant crown 2 days later. Sutures are removed 1 week after the surgery.
  Arms: Scarf connective tissue graft
Procedure: Dual zone concept after immediate implant placement — DBBM is applied and condensed up to the level of the buccal soft tissue margin. A healing abutment is installed, which is replaced by a provisional implant crown 2 days later. Usually, sutures are not needed in this group, unless minimal papilla opening was required to extract the tooth. In that case, sutures will be removed after 1 week.
  Arms: Dual zone concept

SUMMARY:
Patients undergoing single immediate implant placement (IIP) in the premaxilla will be invited to participate in this randomized controlled trial (RCT). Prior to surgery, a small- field low-dose cone beam computed tomography (CBCT) is taken to verify the integrity of the facial bone wall and an adequate amount of apical and palatal bone availability for implant anchorage. 54 patients will be randomly assigned to either conventional connective tissue graft (C-CTG), scarf tissue graft (S-CTG) or dual zonde conept (DZ). Sealed envelopes are prepared for that purpose, of which 18 are internally labeled as C-CTG, 18 as S-CTG and 18 as DZ. Following IIP, a sealed envelope will be opened to reveal the treatment concept.

Successful regeneration (primary outcome) is achieved when the combination of socket grafting and transmucosal augmentation (C-CTG or S-CTG or DZ) would be able to counteract any buccal soft tissue loss at level -1 mm. It is assessed on the basis of superimposed CBCTs taken pre-operatively and at one-year follow-up. Secondary outcomes include: horizontal buccal bone loss, vertical buccal bone loss, increase in buccal soft tissue thickness, patient-reported outcomes, plaque, bleeding on probing, probing depth, marginal bone loss, change in buccal soft tissue profile, midfacial soft tissue level, mesial and distal papilla level, Pink Esthetic Score.

DETAILED DESCRIPTION:
This study is a three-arm randomized controlled trial comparing conventional connective tissue grafting (C-CTG) with two alternative soft-tissue augmentation approaches-scarf CTG (S-CTG) and the dual-zone technique (DZ)-in patients receiving single immediate implant placement in the anterior maxilla. The primary objective is to determine which method results in the highest proportion of sites showing successful regeneration 1 mm below the implant shoulder. Secondary outcomes assess clinical parameters, patient-reported pain and medication use, hard- and soft-tissue dimensional changes, and esthetic scores.

Eligible participants are adults with good oral hygiene and an anterior maxillary tooth requiring extraction with adequate bone support. Exclusion criteria include pregnancy, systemic disease, smoking, active infection, periodontal disease, and extensive gingival asymmetry. Fifty-four patients will be randomized equally to the three intervention groups; allocation is concealed and outcome assessors are blinded.

All patients receive immediate implant placement with socket grafting. The three groups differ only in the soft-tissue augmentation method: C-CTG involves placing a connective tissue graft in a buccal pouch; S-CTG uses a smaller graft fixed at the transmucosal aspect without a pouch; DZ relies on graft condensation beneath the soft tissue without a connective tissue graft. Standard postoperative care is provided in all groups.

Hard- and soft-tissue changes are assessed using cone-beam CT, clinical measurements, intra-oral scans, and standardized photography at baseline and follow-up visits. Successful regeneration is defined by maintenance of buccal soft tissue at the specified reference level. Patient-reported postoperative pain and analgesic use are recorded after one week. Esthetic outcomes are evaluated using a validated scoring system at 1- and 5-year follow-up.

Data will be analyzed using appropriate statistical tests for group comparisons, including mixed models for tissue changes, Fisher's exact test for the primary outcome, and non-parametric tests for variables that are not normally distributed. A two-sided significance level of 5% is applied throughout.

ELIGIBILITY:
Inclusion Criteria:

* At least 20 years old
* Good oral hygiene defined as full-mouth plaque score ≤ 25%
* Presence of an incisor, cuspid or premolar in the maxilla that needs to be extracted for any reason with at least one neighboring tooth present
* At least 3 mm bone available at the apical or palatal aspect of the alveolus as assessed on CBCT to ensure primary implant stability
* Intact buccal bone wall (type I) or limited buccal bone dehiscence (type IIa or IIb) at the time of extraction
* Written informed consent.

Exclusion Criteria:

* Pregnancy
* Systemic diseases
* Smoking; suppuration
* > 1 mm gingival asymmetry between the failing and contralateral tooth
* Untreated periodontal disease
* Untreated caries lesions.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2031-11-01 (Estimated)

PRIMARY OUTCOMES:
Succesful regeneration (%) | 1-, 5 year
  Successful regeneration is achieved when the combination of socket grafting and transmucosal augmentation (C-CTG or S-CTG or DZ) would be able to counteract any buccal soft tissue loss at level -1 mm. It is assessed on the basis of superimposed CBCTs taken pre-operatively and at one-year follow-up.

SECONDARY OUTCOMES:
Horizontal buccal bone loss -1, -3 and -5 (mm) | 1-, 5 year
  Horizontal buccal bone loss at level -1 mm is calculated by subtracting the pre-operative horizontal buccal bone level from the 1-year horizontal buccal bone level, both at level -1 mm. Hence, negative values represent bone loss. The same methodology is applied to determine horizontal buccal bone loss at level -3 and -5 mm.
Vertical bone loss (mm) | 1-, 5 year
  Vertical buccal bone level is measured as the vertical distance from the buccal bone peak to the reference line at the level of the implant-abutment interface to the nearest 0.1 mm. Vertical buccal bone loss is calculated by subtracting the pre-operative vertical bone level from the 1-year vertical bone level. Hence, negative values represent bone loss.
Increase in buccal soft tissue thickness (mm) | 1-, 5 year
  Buccal soft tissue thickness is measured as the distance from the buccal bone surface to the buccal soft tissue profile at level -1 mm to the nearest 0.1 mm. Increase in buccal soft tissue thickness is calculated by subtracting its pre-operative value from the 1-year value. Hence, positive values represent tissue gain.
Patient-reported outcomes | 1-, 5 year
  One week after surgery, patients will be asked how many analgesics have been taken. In addition, they will be asked to rate postoperative pain on a numeric rating scale (0-10).
Plaque (%) | 1-, 5 year
  At 1-year and 5-year follow-up the treating surgeon evaluates plaque at four sites around the implant (mesial, buccal, distal, palatal). Each area receives a score of 0 or 1, representing the absence or presence of plaque.
Bleeding on probing (%) | 1-, 5 year
  At 1-year and 5-year follow-up the treating surgeon evaluates bleeding on probing at four sites around the implant (mesial, buccal, distal, palatal). Each area receives a score of 0 or 1, representing the absence or presence of bleeding on probing.
Probing depth (mm) | 1-, 5 year
  At 1-year and 5-year follow-up the treating surgeon evaluates probing depth at four sites around the implant (mesial, buccal, distal, palatal). Probing depth is registered with a manual probe (University North Carolina Probe PCPUNC 156, Hu-Friedy, Frankfurt, Germany) and measurements are rounded up to the nearest 0.5 mm. A mean value is calculated per implant.
Marginal bone loss (mm) | 1-, 5 year
  Changes in the distance from the implant-abutment interface to the first bone-to-implant contact (so-called marginal bone level) at the mesial and distal aspect of each implant as measured on 2D intra-oral radiographs.
Change in buccal soft tissue profile (mm) | 1-, 5 year
  Changes in buccal soft tissue profile as measured on superimposed digital surface models. An intra-oral scan is taken prior to implant surgery and at 1- and 5- year follow up. On the obtained digital models, an area of interest (AOI) at the buccal aspect was drawn for each site. The AOI extends from 0.5 mm below the soft tissue margin to 4 mm more apical. In mesio-distal dimension, the AOI reaches from the mesial to the distal line angle. The AOI may vary between sites because of individual anatomic differences but must be kept constant in each site across time points. A volumetric change (mm3) was calculated by designated software within the AOI and divided by the AOI surface (mm2). This results in the mean change in buccal soft tissue profile (mm).
Change in midfacial soft tissue level (mm) | 1-, 5 year
  Change in midfacial soft tissue level from surgery to 1-year and 5-year follow-up is calculated on digital surface models from in the same software (SMOP, Swissmeda AG, Zurich, Switzerland). First, a reference line is drawn connecting the middle of the incisal edge on both adjacent teeth at both timepoints. Then, the distance from this line to the buccal mucosal margin (so-called midfacial soft tissue level) is determined at the centre of each implant to the nearest 0.01 mm. Change in midfacial soft tissue level is calculated by subtracting midfacial soft tissue level from the preoperative situation from the one at 1-year and 5-year follow-up. Negative values indicate recession; positive values indicate vertical regrowth. Change in midfacial soft tissue level is assessed by a blinded examiner.
Change in mesial and distal papilla level (mm) | 1-, 5 year
  Change in mesial and distal papilla level from surgery to 1-year and 5-year follow-up is calculated at the mesial and distal aspect. The methodology is the same as described for the change in midfacial soft tissue level.
Pink Esthetic Score | 1-, 5 year
  Pink Esthetic Score (PES) is registered by a trained and blinded examiner using frontal and occlusal clinical pictures taken at 1 year and 5-year follow-up. The PES results in a score from 0 (worst esthetic outcome) to 14 (perfect esthetic outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- Ghent University Hospital, Ghent, East Flanders, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
If the data can be included in a meta-analysis upon request by the authors, they can be transferred

REFERENCES:
- [Background] Zuiderveld EG, van Nimwegen WG, Meijer HJA, Jung RE, Muhlemann S, Vissink A, Raghoebar GM. Effect of connective tissue grafting on buccal bone changes based on cone beam computed tomography scans in the esthetic zone of single immediate implants: A 1-year randomized controlled trial. J Periodontol. 2021 Apr;92(4):553-561. doi: 10.1002/JPER.20-0217. Epub 2020 Sep 11. PMID 32918332
- [Background] Wanis RW, Hosny MM, ElNahass H. Clinical evaluation of the buccal aspect around immediate implant using dual zone therapeutic concept versus buccal gap fill to bone level: A randomized controlled clinical trial. Clin Implant Dent Relat Res. 2022 Jun;24(3):307-319. doi: 10.1111/cid.13091. Epub 2022 May 4. PMID 35507735
- [Background] Tonetti MS, Jung RE, Avila-Ortiz G, Blanco J, Cosyn J, Fickl S, Figuero E, Goldstein M, Graziani F, Madianos P, Molina A, Nart J, Salvi GE, Sanz-Martin I, Thoma D, Van Assche N, Vignoletti F. Management of the extraction socket and timing of implant placement: Consensus report and clinical recommendations of group 3 of the XV European Workshop in Periodontology. J Clin Periodontol. 2019 Jun;46 Suppl 21:183-194. doi: 10.1111/jcpe.13131. PMID 31215112
- [Background] Slagter KW, Meijer HJA, Hentenaar DFM, Vissink A, Raghoebar GM. Immediate single-tooth implant placement with simultaneous bone augmentation versus delayed implant placement after alveolar ridge preservation in bony defect sites in the esthetic region: A 5-year randomized controlled trial. J Periodontol. 2021 Dec;92(12):1738-1748. doi: 10.1002/JPER.20-0845. Epub 2021 Apr 3. PMID 33724473
- [Background] Sicilia-Felechosa A, Pereira-Fernandez A, Garcia-Lareu J, Bernardo-Gonzalez J, Sicilia-Blanco P, Cuesta-Fernandez I. Flapless immediate implant placement and provisionalization in periodontal patients: A retrospective consecutive case-series study of single-tooth sites with dehiscence-type osseous defects. Clin Oral Implants Res. 2020 Mar;31(3):229-238. doi: 10.1111/clr.13559. Epub 2020 Jan 20. PMID 31755601
- [Background] Seyssens L, Eghbali A, Cosyn J. A 10-year prospective study on single immediate implants. J Clin Periodontol. 2020 Oct;47(10):1248-1258. doi: 10.1111/jcpe.13352. Epub 2020 Sep 2. PMID 32748983
- [Background] Seyssens L, Eeckhout C, Cosyn J. Immediate implant placement with or without socket grafting: A systematic review and meta-analysis. Clin Implant Dent Relat Res. 2022 Jun;24(3):339-351. doi: 10.1111/cid.13079. Epub 2022 Mar 21. PMID 35313067
- [Background] Seyssens L, De Lat L, Cosyn J. Immediate implant placement with or without connective tissue graft: A systematic review and meta-analysis. J Clin Periodontol. 2021 Feb;48(2):284-301. doi: 10.1111/jcpe.13397. Epub 2020 Nov 20. PMID 33125754
- [Background] Raghoebar GM, Korfage A, Meijer HJA, Gareb B, Vissink A, Delli K. Linear and profilometric changes of the mucosa following soft tissue augmentation in the zone of aesthetic priority: A systematic review and meta-analysis. Clin Oral Implants Res. 2021 Oct;32 Suppl 21:138-156. doi: 10.1111/clr.13759. PMID 34642988
- [Background] O'Leary TJ, Drake RB, Naylor JE. The plaque control record. J Periodontol. 1972 Jan;43(1):38. doi: 10.1902/jop.1972.43.1.38. No abstract available. PMID 4500182
- [Background] Mareque S, Castelo-Baz P, Lopez-Malla J, Blanco J, Nart J, Valles C. Clinical and esthetic outcomes of immediate implant placement compared to alveolar ridge preservation: a systematic review and meta-analysis. Clin Oral Investig. 2021 Aug;25(8):4735-4748. doi: 10.1007/s00784-021-03986-6. Epub 2021 Jun 7. PMID 34100157
- [Background] Kan JYK, Yin S, Rungcharassaeng K, Zucchelli G, Urban I, Lozada J. Facial implant gingival level and thickness changes following maxillary anterior immediate tooth replacement with scarf-connective tissue graft: A 4-13-year retrospective study. J Esthet Restor Dent. 2023 Jan;35(1):138-147. doi: 10.1111/jerd.12996. Epub 2022 Dec 13. PMID 36511151
- [Background] Griffin TJ, Cheung WS, Zavras AI, Damoulis PD. Postoperative complications following gingival augmentation procedures. J Periodontol. 2006 Dec;77(12):2070-9. doi: 10.1902/jop.2006.050296. PMID 17209793
- [Background] Furhauser R, Florescu D, Benesch T, Haas R, Mailath G, Watzek G. Evaluation of soft tissue around single-tooth implant crowns: the pink esthetic score. Clin Oral Implants Res. 2005 Dec;16(6):639-44. doi: 10.1111/j.1600-0501.2005.01193.x. PMID 16307569
- [Background] Fettouh AIA, Ghallab NA, Mina NA, Abdelmalak MS, Abdelrahman AAG, Shalaby AF, Shemais N. Hard and soft tissue alterations using dual-zone concept versus connective tissue graft at maxillary immediate implant placement: A 1-year randomized clinical and volumetric trial. Clin Oral Implants Res. 2024 May;35(5):510-525. doi: 10.1111/clr.14247. Epub 2024 Feb 19. PMID 38372450
- [Background] Elaskary A, Ghallab N, Thabet A, Shemais N. The bone shielding versus dual-zone concept in treating thin-walled fresh extraction sockets with immediate implant placement: Soft and hard tissue changes. A randomized clinical trial. Clin Implant Dent Relat Res. 2024 Feb;26(1):66-77. doi: 10.1111/cid.13275. Epub 2023 Sep 5. PMID 37669913
- [Background] Cosyn J, Struys T, Van Hove PJ, De Buyser S, De Bruyckere T. A Randomized Controlled Trial on the Timing of Soft-Tissue Augmentation in Immediate Implant Placement: Hard-Tissue Changes and Clinical Outcome. J Clin Periodontol. 2024 Nov;51(11):1534-1544. doi: 10.1111/jcpe.14060. Epub 2024 Sep 1. PMID 39218777
- [Background] Cosyn J, De Lat L, Seyssens L, Doornewaard R, Deschepper E, Vervaeke S. The effectiveness of immediate implant placement for single tooth replacement compared to delayed implant placement: A systematic review and meta-analysis. J Clin Periodontol. 2019 Jun;46 Suppl 21:224-241. doi: 10.1111/jcpe.13054. PMID 30624808
- [Background] Chu SJ, Salama MA, Salama H, Garber DA, Saito H, Sarnachiaro GO, Tarnow DP. The dual-zone therapeutic concept of managing immediate implant placement and provisional restoration in anterior extraction sockets. Compend Contin Educ Dent. 2012 Jul-Aug;33(7):524-32, 534. PMID 22908601
- [Background] Botticelli D, Berglundh T, Lindhe J. Hard-tissue alterations following immediate implant placement in extraction sites. J Clin Periodontol. 2004 Oct;31(10):820-8. doi: 10.1111/j.1600-051X.2004.00565.x. PMID 15367183
- [Background] Araujo MG, Sukekava F, Wennstrom JL, Lindhe J. Ridge alterations following implant placement in fresh extraction sockets: an experimental study in the dog. J Clin Periodontol. 2005 Jun;32(6):645-52. doi: 10.1111/j.1600-051X.2005.00726.x. PMID 15882225
- [Background] Assaf JH, Assaf DD, Antoniazzi RP, Osorio LB, Franca FM. Correction of Buccal Dehiscence During Immediate Implant Placement Using the Flapless Technique: A Tomographic Evaluation. J Periodontol. 2017 Feb;88(2):173-180. doi: 10.1902/jop.2016.160276. Epub 2016 Sep 13. PMID 27620655
- See also: FDA (2023) Adjusting for Covariates in Randomized Clinical Trials for Drugs and Biological Products. Guidance for Industry. — https://www.fda.gov/regulatory-information/search-fda-guidance-documents/adjusting-covariates-randomized-clinical-trials-drugs-and-biological-products